CLINICAL TRIAL: NCT06608069
Title: Relationship Between the Variation in Medication Adherence Level and Clinical Outcomes Among Tuberculosis: A Randomized Controlled Trial
Brief Title: Pharmacist-Led Intervention to Improve TB Treatment Adherence
Acronym: RA-15041995
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, AMER HAYAT KHAN, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMRR ID-22-01964-WWH
Record Dates: First submitted 2024-09-03; First posted 2024-09-23 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2024-10

CONDITIONS: Tuberculosis, Pulmonary; HIV Coinfection
MeSH Terms: conditions — Tuberculosis, Pulmonary; HIV Infections

STUDY DESIGN:
Intervention Model Description: The goal of this clinical trial is to compare the adherence of co-morbid patients in control and experimental group
  The main question[s]it aims to answer are:
  * How will pharmacist-led interventions improve the medication adherence level of TB and HIV con-infected patients?
  * Has there been an increase in the adherence level of co-infected patients following pharmacist-led interventions?
  Participants will be interviewed to measure the level of adherence.
  If there is a comparison group:
  Enrolled patient will be counselled and educated by pharmacist on the therapy and benefits of adherence (Control group).
  Enrolled participants will be counselled and educated by pharmacist on the therapy and benefits of adherence. Patients will be reminded to take the medication through SMS every day by the pharmacist (Experimental group).
Masking Description: To ensure the security of the patients' information, a double-blind randomization technique will be adopted. The computer gives each patient a code number, and the code numbers will then be allocated randomly to the treatment groups. All data will be kept in a database, and backup file with password protectors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational councelling and Reminder. (Experimental): Enrolled participants will be counselled and educated by pharmacist on the therapy and benefits of adherence.
  Interventions: Behavioral: Educational counselling
- DOTS therapy (No Intervention): Enrolled patient will be given the DOT therapy for TB.

INTERVENTIONS:
Behavioral: Educational counselling — Enrolled participants will be counselled and educated by pharmacist on the therapy and benefits of adherence.
  Arms: Educational councelling and Reminder.

SUMMARY:
The goal of this clinical trial is to compare the adherence of co-morbid patients in control and experimental group

The main question[s]it aims to answer are:

1. To evaluate the impact of pharmacist-led educational intervention on treatment adherence among patients with PTB using the health belief model theory and MARS-5.
2. To evaluate the impact of pharmacist-led educational intervention on treatment outcomes among patients with PTB.
3. To evaluate the impact of pharmacist-led educational intervention on HRQoL among patients with PTB.

Participants will be interviewed to measure the level of adherence.

If there is a comparison group:

The enrolled patient will be counselled and educated by the pharmacist on the therapy and the benefits of adherence (Control group).

Enrolled participants will be counselled and educated by pharmacist on the therapy and benefits of adherence. (Experimental group).

DETAILED DESCRIPTION:
In 2019, tuberculosis (TB) remained the leading cause of death due to a single infectious pathogen. An estimated 10 million people had TB worldwide, with 1.2 million TB fatalities among Human immune deficiency virus (HIV)-negative people and 208, 000 deaths among HIV-positive people. Literature indicated that treatment adherence for coinfections diseases is difficult due to the complexity, low tolerability, and extended duration of current treatment regimens, especially for both drug-susceptible and drug-resistant TB. There is a need for continuing the quest for low-cost, reliable, and acceptable measures of adherence for the treatment of TB and HIV co-infection. A qualitative approach and pharmacist-led intervention are needed to improve the adherence level of medication for TB patients. The study is aimed to investigate the degree of adherence and evaluate its impacts on clinical outcomes in TB and HIV co-infected patients. To determine the uptake and usage of the intervention, the study will include nested qualitative and economic evaluation sub-studies as well as a process evaluation. A longitudinal study design will adopt to carry out the present study, involving TB and HIV co-infected patients in either the pharmacist-led intervention (adherence and medication reminder, follow-up reminders, and counselling) or control arm. To determine the uptake and usage of the intervention, the study will include theoretical and conceptual models and theories. The study will conclude with targeted efforts of Pharmacist led intervention to improve and sustain excellent adherence in the real-world clinical setting which is critical for maximizing the effectiveness of each medication and treatment. These innovative technologies can thereby be harnessed to improve adherence to TB and HIV regimens in Malaysia and worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or more.
* Newly bacteriologically confirmed TB case.

Exclusion Criteria:

* Pregnancy and any medical condition unrelated to TB

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Level of adherence among PTB patients. | 6 months
  The patient's level of adherence will be checked using the Health Belief Model Questionnaire and the MARS-5 adherence scale, as well as the patient's interview. The MARS-5 scores will indicate if a patient is adherent or not. Scores are calculated as, Score individual items (5 = never to 1 = always) i.e. high scores = high adherence.
  Add the individual scores to form a scale score (range = 5 to 25).

CONTACTS AND LOCATIONS:
Overall Officials: Aner H Khan, Principal Investigator — Universiti Sains Malaysia
Locations (2):
- Malaysia (2):
  - Hospital Pulau Pinang, George Town
  - Universiti Sains Malaysia, George Town

IPD SHARING:
Plan to Share IPD: No